CLINICAL TRIAL: NCT00351611
Title: PROSPECTIVE RANDOMIZED 12-WEEK CONTROLLED STUDY OF VISUAL FIELD CHANGE IN SUBJECTS WITH PARTIAL SEIZURES RECEIVING PREGABALIN OR PLACEBO
Brief Title: Vision Testing in Patients With Partial Seizures Receiving Either Lyrica or Placebo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: A0081096; 2009-014269-25 (EudraCT Number)
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Epilepsies, Partial
Keywords: epilepsy partial seizure treatment with pregabalin or placebo; vision testing
MeSH Terms: conditions — Epilepsies, Partial | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active drug
  Interventions: Drug: Lyrica (pregabalin)
- Placebo (Placebo Comparator): placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lyrica (pregabalin) — 150 mg twice a day, oral administration
  Arms: Active
Drug: placebo — Twice a day, oral administration
  Arms: Placebo

SUMMARY:
Patients with partial seizures currently taking 1-3 antiepileptic medications will have a 50:50 chance to receive Lyrica 300 mg per day or placebo (no active ingredients) added on to their current medications for 3 months. Neither the study doctor nor the patient will know the medication assignment. Vision testing will be performed prior to receiving the study treatment and at the end of the study to see if there are any changes.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy partial seizure subjects.
* Currently taking 1 to 3 antiepileptic drugs.

Exclusion Criteria:

* Pre-existing eye diseases (glaucoma).
* Insufficient response to pregabalin in the treatment of partial seizure, or patients currently receiving pregabalin treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2006-07-26 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (149):
- United States (102):
  - Neurology Center, P.C., Mobile, Alabama
  - Premier Medical Group, Mobile, Alabama
  - Neurology Clinic, PC, Northport, Alabama
  - North River Ophthalmology, Tuscaloosa, Alabama
  - Western Neurosurgery, Tucson, Arizona
  - Office of Robert Snyder, MD, Tucson, Arizona
  - REM Medical Clinical Research, Tucson, Arizona
  - NEA Baptist Clinic - Clinical Research Center, Jonesboro, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - NEA Baptst Clinic, Jonesboro, Arkansas
  - Chenal MRI, Little Rock, Arkansas
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Eye Care Arkansas, Little Rock, Arkansas
  - Radiology Consultants, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Barbara Swartz, MD, Inc, Costa Mesa, California
  - Mireille P. Hamparian, Glendale, California
  - Lakeside Vision Center, Irvine, California
  - Eye Treatment Center, Inc., Long Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Clinical Innovations, Inc., Paramount, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Bradenton Research Center, Inc, Bradenton, Florida
  - The Eye Associates, Bradenton, Florida
  - SJS Clinical Research, Inc., Destin, Florida
  - White Wilson Medical Center, Fort Walton Beach, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Dr. Raul F. Masvidal, MD, PA, Miami, Florida
  - David M Klein, MD, PA, Port Charlotte, Florida
  - Medsol Clinical Research Center, Inc, Port Charlotte, Florida
  - Intercoastal Medical Research Center, Sarasota, Florida
  - Dr. Nicholas Monsul, Sarasota, Florida
  - Sarasota Retinal Institute, Sarasota, Florida
  - Coastal Research Associates, LLC, Atlanta, Georgia
  - Comprehensive Neurology Specialists, PC, Suwanee, Georgia
  - Professional Research Network of Kansas, Wichita, Kansas
  - Vitreo-Retinal Consultants and Surgeons, Wichita, Kansas
  - Neuromedical Clinic of Central Louisiana, Alexandria, Louisiana
  - Louisiana Eye and Laser Center, Alexandria, Louisiana
  - University of Maryland Eye Associates, P.A., Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Glaucoma Plus Eye Care, LLC, Columbia, Maryland
  - Center for Brain and Neuro Care, LLC, Fulton, Maryland
  - Bergman Eye Associates, Hagerstown, Maryland
  - Neurology Consultant, P.A., Hagerstown, Maryland
  - The Center for Clinical Research, Hagerstown, Maryland
  - Harper Hospital, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Fraser Eye Care Center, Fraser, Michigan
  - Minneapolis Clinic of Neurology, Ltd, Golden Valley, Minnesota
  - University of Missouri, Columbia, Missouri
  - CCN-MS & Neurology Associates, Columbia, Missouri
  - Nevada Eye Care, Las Vegas, Nevada
  - Neurology Center of Las Vegas, Las Vegas, Nevada
  - Institute of Neurological Care, Englewood Cliffs, New Jersey
  - Office of Patricia Burke, MD, Paramus, New Jersey
  - Dent Neurologic Institute, Amherst, New York
  - Dent Neurosciences Research Center, Amherst, New York
  - Western New York Ophthalmology Group, Amherst, New York
  - Buffalo General Hospital, Buffalo, New York
  - The Jacobs Neurological Institute Comprehensive Epilepsy Center, Buffalo, New York
  - Guilford Neurologic Associates, Inc, Greensboro, North Carolina
  - Digby Eye Associates, Greensboro, North Carolina
  - Clinical Research of Winston-Salem, Winston-Salem, North Carolina
  - Salem Neurological Center, PA, Winston-Salem, North Carolina
  - Office of Dr. James D. Branch, MD, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - The Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Jeffrey Shaver, MD, Edmond, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Clinical Trials of America, Inc., Eugene, Oregon
  - Oregon Eye Consultants, LLC, Eugene, Oregon
  - Pacific Women's Center, LLC, Eugene, Oregon
  - Oregon Neurology Associates, Springfield, Oregon
  - Daniel J. Nadler, MD, PC, Beaver, Pennsylvania
  - Heritage Valley Health System, Beaver, Pennsylvania
  - Valley Neurological Associates, Monaca, Pennsylvania
  - Center For Advanced Eye Care, Greenville, South Carolina
  - Premier Neurology, PC, Greer, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Glaucoma Consultants and Center for Eye Research, PA, Mt. Pleasant, South Carolina
  - Tidewater Neurology, Mt. Pleasant, South Carolina
  - Neurology Centers of the Carolinas, Spartanburg, South Carolina
  - Piedmont Eye Associates, Spartanburg, South Carolina
  - Envision Eye Care, Bristol, Tennessee
  - Tri-state Mountain Neurology Associates, PC, Johnson City, Tennessee
  - Semmes Murphey Clinic, Memphis, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Texan Eye, Austin, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Glaucoma Associates of Texas, Dallas, Texas
  - Egret Bay Neurology, PA, Houston, Texas
  - DeHaven Eye Clinic, Longview, Texas
  - Diagnostic Clinic of Longview Center for Clinical Research, Longview, Texas
  - Diagnostic Clinic of Longview, PA, Longview, Texas
  - Coastal Eye Associates, Webster, Texas
  - Neurological Associates Sarah Cannon Cancer Institute;, Richmond, Virginia
  - Medical College of Wisconsin Department of Neurology Froedtert Memorial Hospital, Milwaukee, Wisconsin
  - Medical College of Wisconsin Eye Institute, Milwaukee, Wisconsin
- Bulgaria (6):
  - DKC 2, Sofia
  - Chetvarta nevrologichna klinika, Sofia
  - Otdelenie po Nevrologia, Vtora MBAL, Sofia
  - Otdelenie po nevrologia, MBAL "Tokuda Bolnitsa", Sofia
  - Universitetska mnogoprofilna bolnitsa za aktivno lechenieAleksandrovska, Klinika po Nevrologia, Sofia
  - Otdelenie po nervni bolesti, MBAL Doverie, Sofia
- Czechia (3):
  - Fakultni Thomayerova nemocnice, Prague
  - NEUROPS s.r.o., Rychnov nad Kněžnou
  - Ocni ambulance, Rychnov nad Kněžnou
- Hungary (5):
  - Synexus Kft., Budapest
  - Budapest Retina Associates Kft., Budapest
  - Orszagos Idegtudomanyi Intezet, Stroke es Epilepszia Osztaly, Budapest
  - Orszagos Idegtudomanyi Intezet, Budapest
  - Csongrad Megyei Egeszsegugyi Ellato Kozpont Hodmezovasarhely-Mako,, Hódmezővásárhely
- India (17):
  - Netra Diagnostics (P) Ltd, Abids, Hyderabad, Andhra Pradesh
  - Krishna Institute of Medical Sciences Ltd., Secunderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - St. John's Medical College Hospital, Bangalore, Karnataka
  - M.S. Ramaiah Medical College and Hospitals,, Bangalore, Karnataka
  - Mallikatta Neuro Center, Mangalore, Karnataka
  - Kasturba Medical College and Hospital,, Manipal, Karnataka
  - Eye Site,, Indore, Madhya Pradesh
  - M.G.M. Medical College & M. Y. Hospitals,, Indore, Madhya Pradesh
  - T.N.M.C and B.Y.L Nair Charitable Hospital,, Mumbai, Maharashtra
  - Kelkar Nursing Home, Pune, Maharashtra
  - Sahyadri Clinical Research Development Centre, A unit of Sahyadri Hospitals Ltd,, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Vijaya Health Centre, Chennai, Tamil Nadu
  - Yashoda Hospital, Hyderabad, Telangana
  - Dr. Ram Manohar Lohia Hospital, New Delhi
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Mexico (3):
  - Instituto Biomedico de Investigacion AC, Aguascalientes, Aquascalientes
  - Dr. Ruben Munoz Flores de la Torre Ophthalmic Office, Aquascalientes, Aquascalientes
  - Hospital Central Dr. Ignacio Morones Prieto, San Luis Potosí City
- Poland (6):
  - Niepubliczny Zaklad Opieki Zdrowotnej "OKOmed" s.c., Goczałkowice Zdrój
  - NZOZ Tommed, Katowice
  - Centrum Medyczne Dendryt, Katowice
  - Prywatny Gabinet Psychiatryczny dr Ewa Dereszak-Kozanecka, Krakow
  - Prywatny Gabinet Okulistyczny dr. n.med. Teresa Gedliczka, Krakow
  - NZOZ Centrum Leczenia Padaczki i Migreny, Krakow
- South Korea (5):
  - Keimyung University Dongsan Hospital, Daegu
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Thailand (2):
  - Khon Kaen University, Faculty of Medicine, Neurology Unit, Department of Medicine, Muang, Changwat Khon Kaen
  - Phramongkutklao hospital,, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081096&StudyName=Vision%20Testing%20in%20Patients%20with%20Partial%20Seizures%20Receiving%20Either%20Lyrica%20or%20%20Placebo

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Participants were randomized to receive pregabalin. In Week 1 (titration), participants received pregabalin 150 milligram per day (mg/day) as 75 mg oral capsules twice daily. From Week 2 to 12, participants received pregabalin 300 mg/day as 150 mg oral capsules twice daily. In Week 13 (tapering), participants received 150 mg/day as 75 mg oral capsules twice daily. Participants were followed up from Week 14 to 15. If participants not tolerated 300 mg/day dose, they were discontinued from the study.
- Placebo: Participants were randomized to receive placebo matched to pregabalin from Week 1 to 13 and were followed up from Week 14 to 15.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 89 | 98
Treated | 89 | 98
Completed | 75 | 88
Not Completed | 14 | 10
Not completed — Adverse Event | 11 | 3
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — No Longer Willing to Participate in Study | 0 | 5
Not completed — Other | 1 | 0
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants randomized to treatment, who received at least 1 dose of study medication.
Groups:
- Pregabalin: Participants were randomized to receive pregabalin. In Week 1 (titration), participants received pregabalin 150 mg/day as 75 mg oral capsules twice daily. From Week 2 to 12, participants received pregabalin 300 mg/day as 150 mg oral capsules twice daily. In Week 13 (tapering), participants received 150 mg/day as 75 mg oral capsules twice daily. Participants were followed up from Week 14 to 15. If participants not tolerated 300 mg/day dose, they were discontinued from the study.
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 89 | 98 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.1 (12.1) | 39.1 (11.6) | 38.6 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 90
  Male | 45 | 52 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 47 | 51 | 98
  Race: Black | 4 | 5 | 9
  Race: Asian | 34 | 40 | 74
  Race: Others | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Decrease (p<0.05) From Baseline in Threshold Value in Any 5 or More Points in Humphrey 24-2 Swedish Interactive Threshold Algorithm (SITA) Standard Testing at Week 12 or Early Termination
Description: In this primary outcome measure, percentage of participants is reported, with a decrease in the threshold value from baseline to Week 12 or termination in any 5 or more points (in either eye) at the p<0.05 level repeated in the same 5 points on subsequent computerized automated perimetry testing (Humphrey 24-2 SITA standard). It was derived from the Humphrey 24-2 SITA standard visual field analyzer. For each eye there were 52 test points. For each test point, the Humphrey analyzer determined the threshold value for sensitivity to light by the participant. In addition, for each of the 52 points, the test provided probabilities (p<0.05, p<0.02, etc.) that a participant with normal vision of the same age would have the same result, i.e., that the measured value at that point was at or below the respective percentile of the age-specific empiric distribution at that position of the field for normal participants.
Time Frame: Baseline, Week 12 or Early Termination (any time up to Week 12)
Population: Per protocol population included all participants randomized to treatment who received at least 1 dose of study medication and excluded participants who had a decrease in at least 5 points at termination but did not return for a repeat test.
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 78 | 90
Percentage of participants | 3.8 | 5.6
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; A 2-sided 95 percent (%) confidence interval (CI) on the difference in percentage of participants, between pregabalin and placebo was constructed using unconditional exact methods; Test type: Non-Inferiority — Non-inferiority was demonstrated if the upper CI bound was less than 0.10 (10%); Difference in percentage of participants = -1.7094, 95% CI 2-sided [-9.1751 to 5.9784]

2. Secondary Outcome: Change From Baseline in Mean Deviation Score From Humphrey Threshold Test at Week 12 or Early Termination
Description: Mean deviation (MD) is a global index of visual field depression. The MD ranges from 0 decibels (no defect) to about -32 decibels (end-stage damage), higher scores indicate worse condition. It is derived from the Humphrey 24-2 SITA standard visual field analyzer. Change in mean deviation score from baseline to Week 12 or termination was computed for each participant. As planned, for each participant, the worst eye (eye with the greatest decrease in mean deviation) was used in the analysis and data is reported for same.
Time Frame: Baseline, Week 12 or Early Termination (any time up to Week 12)
Population: ITT population included all participants randomized to treatment, who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" refers to those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Decibels
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 83 | 96
Decibels | -0.339 (0.1467) | -0.214 (0.1321)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Analysis of covariance (ANCOVA) with treatment and center in the model and the baseline mean deviation as the covariate was used to construct a 2-sided 95% CI on the difference in least squares (LS) mean between pregabalin and placebo; Test type: Non-Inferiority — Non-inferiority with respect to mean deviation was demonstrated if the lower bound of the CI is greater than -2.0 decibels; p = 0.4414, ANCOVA; Difference in LS mean = -0.125, 95% CI 2-sided [-0.443 to 0.194]

3. Secondary Outcome: Change From Baseline in Visual Acuity at Week 12 or Early Termination
Description: Visual acuity best-corrected (with glasses or best possible glasses prescription) was measured using early treatment diabetic retinopathy study (ETDRS) charts. There were 2 ETDRS charts. The letters on chart A were read using the right eye and on chart B using the left eye. The participants started from the top of the chart to down. The participants read down the chart until they reached a row where a minimum of 3 letters on a line could not be read. The participants were scored by number of letters identified correctly. Range was from 0 to 70, with higher scores indicate better visual acuity. As planned, for each participant, the worst eye (eye with the greatest decrease in visual acuity) was used in the analysis and data is reported for same.
Time Frame: Baseline, Week 12 or Early Termination (any time up to Week 12)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Letters identified correctly
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 83 | 94
Letters identified correctly | -1.890 (0.5515) | -0.990 (0.5057)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; ANCOVA with treatment and center in the model and the baseline visual acuity as the covariate was used to construct a 2-sided 95% confidence interval on the difference in LS mean between pregabalin and placebo; Test type: Other; p = 0.1346, ANCOVA; Difference in LS mean = -0.900, 95% CI 2-sided [-2.083 to 0.283]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 15
Description: Same event may appear as both an adverse event and serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety analysis performed on all participants randomized to treatment, who received at least 1 dose of study medication.
Arm/Group | Pregabalin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/89 | 0/98
Serious Adverse Events (participants affected / at risk) | 4/89 | 1/98
Other Adverse Events (participants affected / at risk) | 33/89 | 13/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=89) | Placebo (N=98)
Pneumonia (Infections and infestations) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Postictal state (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=89) | Placebo (N=98)
Fatigue (General disorders) | 6 | 3
Weight increased (Investigations) | 5 | 2
Dizziness (Nervous system disorders) | 20 | 3
Headache (Nervous system disorders) | 3 | 5
Somnolence (Nervous system disorders) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT00351611/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/11/NCT00351611/SAP_001.pdf